CLINICAL TRIAL: NCT04755946
Title: Clinical Study Evaluating the Possible Efficacy and Safety of Roflumilast in Patients With Diabetic Nephropathy
Brief Title: Possible Role of Roflumilast in Diabetic Nephropathy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Hisham Mohammad Abd-El-Galil El-Nahhas, Pharm D, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Roflumilast in DN
Record Dates: First submitted 2021-02-13; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Diabetic Nephropathies
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- roflumilast arm (Experimental)
  Interventions: Drug: Roflumilast
- placebo arm (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roflumilast — adding one tablet of roflumilast 500 mcg to the standard ACEI (captopril) for diabetic nephropathy management
  Arms: roflumilast arm
Drug: Placebo — Placebo
  Arms: placebo arm

SUMMARY:
adding roflumilast to the standard therapy for diabetic nephropathy and studying the progression of many outcomes including urinary albumin to creatinine ratio, estimated GFR, biomarkers of diabetic nephropathy

ELIGIBILITY:
Inclusion Criteria: diabetic patients with persistent micro- or macroalbuminuria despite treatment with the maximum tolerated dose of ACE inhibitors for at least 8 weeks before the screening and randomization

* Type I or II diabetic patient with stage 2 CKD (eGFR = 60 - 89 ml/min) ,stage 3 CKD (eGFR = 30 - 59 ml/min) or stage 4 (eGFR 15-29 ml/min)

Exclusion Criteria:

* moderate to severe hepatic disease (Child-Pugh B or C) severe renal disease (eGFR<15 ml/min) body-mass index below 25 kg/m2 concomitant use of strong cytochrome P450 inducers (e.g. rifampicin, phenobarbital, carbamazepine, phenytoin) known psychiatric illness, congestive heart disease patients with allergy for roflumilast pregnant and lactating women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-03-10 (Estimated); Primary Completion 2021-06-10 (Estimated); Study Completion 2021-07-10 (Estimated)

PRIMARY OUTCOMES:
Percent change in urinary albumin creatinine ratio (UACR) | Baseline and 3 months
  measuring UACR pre and post experiment and substracting and dividing on baseline level
Absolute change in Estimated glomerular filtration rate (eGFR) | Baseline and 3 months
  substracting pre-treatment from post-treatment values of EGFR

SECONDARY OUTCOMES:
Change in Urinary pro-inflammatory cytokine MCP-1 | Baseline and 3 months
  substracting pre-treatment from post-treatment values of Change in Urinary pro-inflammatory cytokine MCP-1
Change in serum irisin level | Baseline and 3 months
  substracting pre-treatment from post-treatment values of serum irisin level

CONTACTS AND LOCATIONS:
Overall Officials: Hisham M Elnahhas, Pharm D, Principal Investigator — Pharm D

IPD SHARING:
Plan to Share IPD: No
data of outcomes and other research but not personal data are intended to be published in application to scientific journals